CLINICAL TRIAL: NCT01926093
Title: Low Dose Lung CT Scan for Quantitative Analysis in ARDS Patients
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Other Study IDs: Policlinico-08; 3102-28/12/2012
Record Dates: First submitted 2013-08-13; First posted 2013-08-20 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-08

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
Keywords: Acute Respiratory Distress Syndrome (ARDS)
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We aimed to assess the accuracy of visual and quantitative analysis performed on low radiation dose lung CT scan (30-60 mAs)compared with that performed on standard radiation dose lung CT scan (110 mAs), in ARDS patients. If the results in computing lung recruitment will be similar, we will be able to use Low Dose CT scan for monitoring of the evolution of the disease in ARDS patients.

ELIGIBILITY:
Inclusion Criteria:

* Acute Respiratory Distress Syndrome
* CT scan performed for clinical purposes

Exclusion Criteria:

* Age < 18 years
* hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ARDS patients fulfilling the Berlin definition criteria
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Difference between Standard and Low Dose lung CT scan in visual and quantitative analysis | 1 day
  We measured lung recruitment with visual and quantitative analysis both on standard and low dose CT scan.

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, MD, Principal Investigator — IRCCS Ca' Granda - Ospedale MAggiore Policlinico
Locations (1):
- IRCCS Ca' Granda - Ospedale MAggiore Policlinico, Milan, Italy